CLINICAL TRIAL: NCT02970227
Title: Inflammatory Cardiomyopathy Cohort of the SFB/TR19 [Kohorte "Entzündliche Kardiomyopathien" Des Sonderforschungsbereichs/Transregio 19 (SFB/TR19)]
Brief Title: Inflammatory Cardiomyopathy Baseline Cohort (SFB/TR19)
Acronym: SFB/TR19
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: SFB/TR19-001
Record Dates: First submitted 2016-11-09; First posted 2016-11-21 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Cardiomyopathies; Heart Failure
Keywords: heart failure; cardiomyopathies; myocarditis
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Myocarditis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observation — None, observation only

SUMMARY:
cohort of cardiomyopathy patients (suspected or validated inflammatory cardiomyopathy) recruited at baseline by the SFB-TR19 project. Standardized protocols used for the assessment of medical history and examinations, laboratory biomarkers, and the collection of various biosamples for biobanking purposes.

ELIGIBILITY:
Inclusion Criteria:

* suspected inflammatory cardiomyopathy at baseline

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or validated inflammatory cardiomyopathy at baseline
Sampling Method: Non-Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2004-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | 1-year follow-ups
  Hospitalization (HF based. all-cause), interventions (ICD, pacemaker), myocardial infarction

SECONDARY OUTCOMES:
LVEF | 1-year follow-ups
  Left ventricular ejection fraction at time of follow-up
VO2peak | 1-year follow-ups
  Exercise capacity by CPET
QOL | 1-year follow-ups
  Quality of life by questionnaire (Minnesota Living with HF questionnaire)
Mortality | 1-year follow-ups
  Mortality (HF-related, CVD, all-cause)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine B, University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No